CLINICAL TRIAL: NCT02527954
Title: Impact of Y-chromosome Microdeletions From Infertile Men on the Chromosomal Constitution of Their Spermatozoa and Embryos. Combined IntraCytoplasmatic Sperm Injection (ICSI) and Preimplantation Genetic Screening (PGS) as Treatment Strategy.
Brief Title: Aneuploidies in Embryos and Spermatozoa From Patients With Y-chromosome Microdeletions
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Collaborators: IVI Murcia (Other); Igenomix (Industry)
Responsible Party: Principal Investigator, Purificación Hernández, Research Coordinator, Instituto Valenciano de Infertilidad, IVI Alicante
Other Study IDs: 1412-ALC-086-PH
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Male Sterility Due to Y-chromosome Deletions
Keywords: Y-chromosome microdeletions; aneuploidy; embryos; spermatozoa
MeSH Terms: conditions — Male sterility due to Y-chromosome deletions; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood, ejaculated semen or testicular biopsy, blastomere
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infertile with Y-chromosome deletions: No intervention will be performed.
  Couples whose infertile men has a Y-chromosome microdeletion (detected in blood cells by Polymerase chain reaction multiplex) and fulfill the criteria will be included in this group (group 1)
- Infertile without Y-chromosome deletions: No intervention will be performed.
  Couples whose infertile men has not any Y-chromosome microdeletion (detected in blood cells by polymerase chain reaction multiplex) and fulfill the criteria will be included in this group (group 2)

SUMMARY:
In this study, investigators assess, using Fluorescence in situ Hybridization (FISH) and Comparative Genomic Hybridization (CGH) arrays for Preimplantation Genetic Screening (PGS), the incidence of aneuploidies in spermatozoa and embryos from infertile men with and without microdeletions who undergo assisted reproduction in their clinics.

DETAILED DESCRIPTION:
Nowadays, Y-chromosome microdeletions are one of the most common causes of male infertility. With a frequency of 8-20% in non-obstructive azoospermic men and 3-14% in severe oligozoospermic men, is the most usual chromosome anomaly associated with failure in sperm production, although the frequency seems to change due to differences in the experimental designs, the ethnic differences, the genetic background, or even environmental influences.

The absence of some genes located on certain regions in the long arm of the human Y chromosome, known as the azoospermia factor region (AZF), causes spermatogenic failure, while spermatozoa has been found in either the ejaculate or the testicle of most patients. Detection of deletions is crucial for the medical treatment of these patients, since it has a prognostic value in predicting potential success of testicular sperm retrieval in azoospermic patients with certain microdeletions, and allows avoiding invasive techniques in oligozoospermic patients whose sperm production could result in progressive worsening.

The development of assisted reproduction techniques, such as intracytoplasmatic sperm injection (ICSI), together with testicular or epididymis sperm retrieval for azoospermic men has allowed these patients to become fathers using their own gametes. Although the effect of Y-chromosome microdeletions on ICSI outcome is controversial, the ability to vertically transmit that genetic defect, and so the infertility, to the offspring has been accepted. Until recently, no clinical consequences other than infertility were supposed in the ICSI-conceived sons of fathers with deletions. However, different studies in the last years, suggest other potentially risks transmitted to the offspring, such as the development of sexual dysfunction due to sex chromosome abnormalities (Turner or Klinefelter syndromes, etc.) or other somatic disorders with worse health implications caused by chromosome aberrations outside the AZF regions or in autosomes that has been associated to Y-chromosome microdeletions. No major clinical complications than infertility has been described in the offspring born from fathers with deletions to date, but it is important to remember that the first generation of those babies, mainly obtained by ICSI, has just reached maturity. Moreover, the mentioned chromosome anomalies, could stop embryo development or increase miscarriage rate. Few studies focused in the incidence of miscarriages in these couples but microdeletions have been detected more frequents in men from couples with recurrent pregnancy loss.

In order to offer fully genetic counseling to these couples, further studies focusing on the relationship between Y-chromosome microdeletions and other chromosomal abnormalities, which also provide information about their consequences in their embryos, are required. Thus, the actual risk of transmitting different anomalies associated to microdeletions to those embryos will be clarified, increasing the chances of a successful pregnancy and live birth.

In this study, investigators assess, using Fluorescence in situ Hybridization (FISH) and Comparative Genomic Hybridization (CGH) arrays for Preimplantation Genetic Screening (PGS), the incidence of aneuploidies in spermatozoa and embryos from infertile men with and without microdeletions who undergo assisted reproduction in their clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Couples with male infertility whose man has non-obstructive azoospermia or severe oligozoospermia with ≤5x1000000 spermatozoa/ml.
2. Assisted Reproductive Technology: ICSI with motile spermatozoa and PGS by CGH arrays.
3. Women <38 years if microinjection is carried out in their own eggs, or 38≤ age <50 years if they receive donated eggs.
4. Women with body mass index (BMI)<30.
5. Men<50 years

Exclusion Criteria:

1. Couples with abnormal karyotypes.
2. Women with any uterine pathology or abnormality, hydrosalpinx, thrombophilia or systemic diseases at the time of embryo transfer that could prejudge the outcome of the cycle
3. Couples with repeated miscarriages (≥2) or implantation failures (≥2).
4. Couples whose men has obstructive azoospermia, genital tract infections (mumps, inflammation, varicocele), cryptorchidism, or if he receives any treatment that can reduce the sperm count.
5. Seminal samples processed by Magnetic Activated Cell Sorting (MACS) technique.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples undergoing "In vitro" Fertilization (IVF) treatment whose man has non-obstructive azoospermia or severe oligozoospermia (≤ 5x1000000 spermatozoa/ml) and consent the genetic analysis of semen samples, as well as the embryo cohort generated by ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-09-22; Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
% Embryos with aneuploidies | three years
  The incidence of embryonic aneuploidies will be examined by CGH arrays analysis after biopsy in day 3 or day 5 of embryo development. This technology allows the analysis of all the chromosomes, so both aneuploidies in gonosomes and autosomes will be determined.
  To measure these percentages the images obtained after CGH array will be analyzed by BlueFuse Software (BlueGnome, Cambridge, UK), identifying normal euploid embryos, embryos with full or partial aneuploidy and chaotic embryos.

SECONDARY OUTCOMES:
% Spermatozoa with aneuploidies | Three years
  The incidence of aneuploidy (%) in sperm will be examined by FISH, analyzing chromosomes 13, 18, 21, X and Y.
  To measure these percentages two examiners will analyze 2000 spermatozoa in each sample.
Fertilization rate (%) | three years
  nº fertilized oocytes/ nº metaphase II oocytes
Day 3 embryos rate (%) | Three years
  nº embryos at day 3/ nº fertilized oocytes
Blastocyst rate (%) | Three years
  nº blastocyst/ nº fertilized oocytes
Cycle efficiency | Four years
  nº transferred embryos + vitrified embryos
Pregnancy rate (%) | Four years
  nº pregnancies/ nº embryos transferred
Biochemical pregnancy rate (%) | Four years
  % of positive pregnancy tests
Clinical pregnancy rate (%) | Four years
  nº pregnancies (proven by the presence of at least 1 embryo with cardiac activity positive by ultrasound after 5-6 weeks of development)/ nº of transfer cycles
Implantation rate (%) | Four years
  nº gestational sacs/ nº transferred embryos
Abortion rate (%) | Four years
  nº miscarriages/ nº pregnancies.
Ongoing pregnancy rate (%) | Four years
  % clinical pregnancies that do not finish in abortion or ectopic pregnancy
Live birth rate (%) | Four years
  Proportion of live birth at home per embryo transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Purificación Hernández-Vargas, PhD, Principal Investigator — Instituto Valenciano de Infertilidad, IVI Alicante
Locations (3):
- Spain (3):
  - IVI Alicante, Alicante
  - IVI Murcia, Murcia
  - Igenomix, Valencia

REFERENCES:
- [Background] Ferlin A, Arredi B, Speltra E, Cazzadore C, Selice R, Garolla A, Lenzi A, Foresta C. Molecular and clinical characterization of Y chromosome microdeletions in infertile men: a 10-year experience in Italy. J Clin Endocrinol Metab. 2007 Mar;92(3):762-70. doi: 10.1210/jc.2006-1981. Epub 2007 Jan 9. PMID 17213277
- [Background] Foresta C, Moro E, Ferlin A. Y chromosome microdeletions and alterations of spermatogenesis. Endocr Rev. 2001 Apr;22(2):226-39. doi: 10.1210/edrv.22.2.0425. PMID 11294825
- [Background] Foresta C, Moro E, Ferlin A. Prognostic value of Y deletion analysis. The role of current methods. Hum Reprod. 2001 Aug;16(8):1543-7. doi: 10.1093/humrep/16.8.1543. PMID 11473940
- [Background] Li Z, Haines CJ, Han Y. "Micro-deletions" of the human Y chromosome and their relationship with male infertility. J Genet Genomics. 2008 Apr;35(4):193-9. doi: 10.1016/S1673-8527(08)60027-2. PMID 18439975
- [Background] Sadeghi-Nejad H, Farrokhi F. Genetics of azoospermia: current knowledge, clinical implications, and future directions. Part II: Y chromosome microdeletions. Urol J. 2007 Fall;4(4):192-206. PMID 18270942
- [Background] Silber SJ. The Y chromosome in the era of intracytoplasmic sperm injection: a personal review. Fertil Steril. 2011 Jun 30;95(8):2439-48.e1-5. doi: 10.1016/j.fertnstert.2011.05.070. PMID 21704208
- [Background] Suganthi R, Vijesh VV, Vandana N, Fathima Ali Benazir J. Y choromosomal microdeletion screening in the workup of male infertility and its current status in India. Int J Fertil Steril. 2014 Jan;7(4):253-66. Epub 2013 Dec 22. PMID 24520494
- [Background] Choi JM, Chung P, Veeck L, Mielnik A, Palermo GD, Schlegel PN. AZF microdeletions of the Y chromosome and in vitro fertilization outcome. Fertil Steril. 2004 Feb;81(2):337-41. doi: 10.1016/j.fertnstert.2003.06.030. PMID 14967370
- [Background] Kihaile PE, Kisanga RE, Aoki K, Kumasako Y, Misumi J, Utsunomiya T. Embryo outcome in Y-chromosome microdeleted infertile males after ICSI. Mol Reprod Dev. 2004 Jun;68(2):176-81. doi: 10.1002/mrd.20074. PMID 15095338
- [Background] Liu XH, Qiao J, Li R, Yan LY, Chen LX. Y chromosome AZFc microdeletion may not affect the outcomes of ICSI for infertile males with fresh ejaculated sperm. J Assist Reprod Genet. 2013 Jun;30(6):813-9. doi: 10.1007/s10815-013-0009-y. Epub 2013 May 30. PMID 23715876
- [Background] Mulhall JP, Reijo R, Alagappan R, Brown L, Page D, Carson R, Oates RD. Azoospermic men with deletion of the DAZ gene cluster are capable of completing spermatogenesis: fertilization, normal embryonic development and pregnancy occur when retrieved testicular spermatozoa are used for intracytoplasmic sperm injection. Hum Reprod. 1997 Mar;12(3):503-8. doi: 10.1093/humrep/12.3.503. PMID 9130751
- [Background] Oates RD, Silber S, Brown LG, Page DC. Clinical characterization of 42 oligospermic or azoospermic men with microdeletion of the AZFc region of the Y chromosome, and of 18 children conceived via ICSI. Hum Reprod. 2002 Nov;17(11):2813-24. doi: 10.1093/humrep/17.11.2813. PMID 12407032
- [Background] Patrat C, Bienvenu T, Janny L, Faure AK, Fauque P, Aknin-Seifer I, Davy C, Thiounn N, Jouannet P, Levy R. Clinical data and parenthood of 63 infertile and Y-microdeleted men. Fertil Steril. 2010 Feb;93(3):822-32. doi: 10.1016/j.fertnstert.2008.10.033. Epub 2008 Dec 4. PMID 19062004
- [Background] Stouffs K, Lissens W, Tournaye H, Van Steirteghem A, Liebaers I. The choice and outcome of the fertility treatment of 38 couples in whom the male partner has a Yq microdeletion. Hum Reprod. 2005 Jul;20(7):1887-96. doi: 10.1093/humrep/deh847. Epub 2005 Mar 24. PMID 15790609
- [Background] van Golde RJ, Wetzels AM, de Graaf R, Tuerlings JH, Braat DD, Kremer JA. Decreased fertilization rate and embryo quality after ICSI in oligozoospermic men with microdeletions in the azoospermia factor c region of the Y chromosome. Hum Reprod. 2001 Feb;16(2):289-92. doi: 10.1093/humrep/16.2.289. PMID 11157822
- [Background] Wu W, Zhou ZM, Lin M, Mao YD, Wang W, Yang XY, Liu JY. [Y-chromosome microdeletions do not affect the outcomes of ICSI for infertile males]. Zhonghua Nan Ke Xue. 2011 Sep;17(9):771-4. Chinese. PMID 21961234
- [Background] Patsalis PC, Sismani C, Quintana-Murci L, Taleb-Bekkouche F, Krausz C, McElreavey K. Effects of transmission of Y chromosome AZFc deletions. Lancet. 2002 Oct 19;360(9341):1222-4. doi: 10.1016/s0140-6736(02)11248-7. PMID 12401251
- [Background] Patsalis PC, Skordis N, Sismani C, Kousoulidou L, Koumbaris G, Eftychi C, Stavrides G, Ioulianos A, Kitsiou-Tzeli S, Galla-Voumvouraki A, Kosmaidou Z, Hadjiathanasiou CG, McElreavey K. Identification of high frequency of Y chromosome deletions in patients with sex chromosome mosaicism and correlation with the clinical phenotype and Y-chromosome instability. Am J Med Genet A. 2005 Jun 1;135(2):145-9. doi: 10.1002/ajmg.a.30712. PMID 15880425
- [Background] Siffroi JP, Le Bourhis C, Krausz C, Barbaux S, Quintana-Murci L, Kanafani S, Rouba H, Bujan L, Bourrouillou G, Seifer I, Boucher D, Fellous M, McElreavey K, Dadoune JP. Sex chromosome mosaicism in males carrying Y chromosome long arm deletions. Hum Reprod. 2000 Dec;15(12):2559-62. doi: 10.1093/humrep/15.12.2559. PMID 11098026
- [Background] Dewan S, Puscheck EE, Coulam CB, Wilcox AJ, Jeyendran RS. Y-chromosome microdeletions and recurrent pregnancy loss. Fertil Steril. 2006 Feb;85(2):441-5. doi: 10.1016/j.fertnstert.2005.08.035. PMID 16595224
- [Background] Jorgez CJ, Weedin JW, Sahin A, Tannour-Louet M, Han S, Bournat JC, Mielnik A, Cheung SW, Nangia AK, Schlegel PN, Lipshultz LI, Lamb DJ. Aberrations in pseudoautosomal regions (PARs) found in infertile men with Y-chromosome microdeletions. J Clin Endocrinol Metab. 2011 Apr;96(4):E674-9. doi: 10.1210/jc.2010-2018. Epub 2011 Jan 20. PMID 21252244
- [Background] Mateu E, Rodrigo L, Martinez MC, Peinado V, Milan M, Gil-Salom M, Martinez-Jabaloyas JM, Remohi J, Pellicer A, Rubio C. Aneuploidies in embryos and spermatozoa from patients with Y chromosome microdeletions. Fertil Steril. 2010 Dec;94(7):2874-7. doi: 10.1016/j.fertnstert.2010.06.046. Epub 2010 Jul 24. PMID 20655521
- [Background] Page DC, Silber S, Brown LG. Men with infertility caused by AZFc deletion can produce sons by intracytoplasmic sperm injection, but are likely to transmit the deletion and infertility. Hum Reprod. 1999 Jul;14(7):1722-6. doi: 10.1093/humrep/14.7.1722. PMID 10402375
- [Background] Perrin A, Douet-Guilbert N, Laudier B, Couet ML, Guerif F, Royere D, Le Bris MJ, De Braekeleer M, Morel F. Meiotic segregation in spermatozoa of a 45,XY,-14,der(18)t(14;18)(q11;p11.3) translocation carrier: a case report. Hum Reprod. 2007 Mar;22(3):729-32. doi: 10.1093/humrep/del420. Epub 2006 Oct 24. PMID 17062581
- [Background] Yogev L, Segal S, Zeharia E, Gamzu R, Maymon BB, Paz G, Botchan A, Hauser R, Yavetz H, Kleiman SE. Sex chromosome alignment at meiosis of azoospermic men with azoospermia factor microdeletion. J Androl. 2004 Jan-Feb;25(1):110-6. doi: 10.1002/j.1939-4640.2004.tb02765.x. PMID 14662793
- [Background] Martinez MC, Bernabe MJ, Gomez E, Ballesteros A, Landeras J, Glover G, Gil-Salom M, Remohi J, Pellicer A. Screening for AZF deletion in a large series of severely impaired spermatogenesis patients. J Androl. 2000 Sep-Oct;21(5):651-5. PMID 10975411
- [Background] Oliva R, Margarit E, Ballesca JL, Carrio A, Sanchez A, Mila M, Jimenez L, Alvarez-Vijande JR, Ballesta F. Prevalence of Y chromosome microdeletions in oligospermic and azoospermic candidates for intracytoplasmic sperm injection. Fertil Steril. 1998 Sep;70(3):506-10. doi: 10.1016/s0015-0282(98)00195-2. PMID 9757880